CLINICAL TRIAL: NCT00315978
Title: Decision Aid to Improve Coronary Heart Disease Risk Modification: a Pilot Randomized Trial
Brief Title: The Impact of Patient Involvement in Decision-Making About Heart Disease Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina (Other)
Organization: University of North Carolina, Chapel Hill (Other)
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: 03-MED-221
Record Dates: First submitted 2006-04-17; First posted 2006-04-19 (Estimated); Last update posted 2007-07-10 (Estimated); Status verified 2006-04

CONDITIONS: Cardiovascular Disease
Keywords: Risk Assessment; Decision Support Technique; Physician-Patient Relations; Prevention and Control
MeSH Terms: conditions — Cardiovascular Diseases

INTERVENTIONS:
Device: Heart-to-Heart Decision Aid

SUMMARY:
The purpose of this study is to determine whether providing patients with information about their global coronary heart disease (CHD) risk and effective risk-reducing strategies allows them to make appropriate decisions about heart disease prevention.

DETAILED DESCRIPTION:
Background: Low utilization of effective CHD prevention strategies may be due to many factors, but chief among them is the lack of patient involvement in prevention decisions. We undertook this study to test the effectiveness of an individually-tailored, computerized decision aid about CHD on patients' discussions with their doctor and their plans for CHD prevention.

Methods: We conducted a pilot randomized trial in a convenience sample of adults with no previous history of cardiovascular disease to test the effectiveness of an individually-tailored, computerized decision aid about CHD prevention against a risk factor list that patients could present to their doctor.

ELIGIBILITY:
Inclusion Criteria:

* presenting for routine medical care with regular medical provider
* able to understand, speak, and read English

Exclusion Criteria:

* prior history of cardiovascular disease
* history of serious medical illness that would limit candidacy for screening
* previous participation in intensive risk modification as part of diabetes study in our clinic
* no cholesterol measurement in the last 3 years, limiting ability to provide up-to-date risk estimate

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2003-06; Study Completion 2004-02

PRIMARY OUTCOMES:
Discussion with provider about CHD risk reduction
Stated plans for CHD risk reduction

SECONDARY OUTCOMES:
Knowledge about CHD prevention
Perception of CHD risk
Interest in participating in decision-making

CONTACTS AND LOCATIONS:
Overall Officials: Stacey L. Sheridan, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Result] Sheridan SL, Shadle J, Simpson RJ Jr, Pignone MP. The impact of a decision aid about heart disease prevention on patients' discussions with their doctor and their plans for prevention: a pilot randomized trial. BMC Health Serv Res. 2006 Sep 27;6:121. doi: 10.1186/1472-6963-6-121. PMID 17005051
- See also: Heart-to-Heart webtool (version 1) tested in research protocol — http://www.med-decisions.com/H2HV2